CLINICAL TRIAL: NCT05616455
Title: Efficacy and Safety of Propionibacterium Extract Gel Versus 0.4% Glyceryl Trinitrate Ointment in the Treatment of Chronic Anal Fissure: a Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Treviso Regional Hospital (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMOR
Record Dates: First submitted 2022-11-05; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Anal Fissure Chronic; Anal Fissure
MeSH Terms: conditions — Fissure in Ano | interventions — chloropentaamminerhodium(III); Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propionibacterium extract gel (Experimental): The Propionibacterium extract gel is a topical product that protect the skin and mucous membranes from external agents. Its film forming property on the epidermis helps reduce inflammation, itching and pain, while the adjunct of antioxidant ingredients helps promote the healing process.
  Patients were instructed to squeeze out from the aluminium tubes containing the Propionibacterium extract gel, 3 grams of gel (3 cm), applying it twice a day for 40 days in the distal anal canal and perianal area.
  Interventions: Drug: Propionibacterium Acnes
- 0.4% glyceryl trinitrate ointment (Active Comparator): 0.4% glyceryl trinitrate ointment is a well-known nitric oxide donor which promotes fissure healing by decreasing resting anal pressure and increasing anoderm blood flow, via the stimulation of the intracellular cyclic GMP resulting in a consequent reduction in cytosolic calcium. The success rate is variable, with 28% of patients experiencing transient headache often leading to drug discontinuation and poor compliance to treatment.
  Patients were instructed to squeeze out from the aluminium tubes containing 0.4% glyceryl trinitrate ointment approximately 1.5 mg of the ointment applying it to the distal anal canal and perianal area with a gloved finger, every 12 hours for 40 days.
  Interventions: Drug: glyceryl trinitrate

INTERVENTIONS:
Drug: Propionibacterium Acnes — Application of the gel every 12 hours for 40 days
  Arms: Propionibacterium extract gel
Drug: glyceryl trinitrate — Application of the gel every 12 hours for 40 days
  Arms: 0.4% glyceryl trinitrate ointment

SUMMARY:
The study compares the efficacy and safety of a Propionibacterium extract gel with 0.4% glyceryl trinitrate ointment in the treatment of chronic anal fissure.

DETAILED DESCRIPTION:
Patients were randomly allocated to a PeG or GTN group and medication was taken every 12 hours for 40 days. Primary outcome was the success rate as measured by a decrease in the REALISE score at 10, 20 and 40 days after starting either treatment. The secondary out-comes were the healing rate, the partial or complete resolution of itching and burning, the rate of complications and adverse events, patients' quality of life and satisfaction at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients diagnosed with chronic anal fissure aged between 18 and 75 years

Exclusion Criteria:

* Fecal incontinence
* Inflammatory bowel disease
* Previous history of anal surgery
* Previous or concomitant treatment for anal fissure, sexually transmitted disease, cancer, immune-suppressive treatment
* Current pregnancy or breastfeeding
* Known allergy to one of the agents contained into the evaluating drugs

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
REALISE score | From baseline to visit 3 (40 days after the start of the treatment)
  REALISE (scoRing systEm for AnaL fIsSurE), was used to assess pain (minimum score = 0, maximum score = 10)

SECONDARY OUTCOMES:
Burning | From baseline to visit 3 (40 days after the start of the treatment)
  Visual analogue scale (VAS) (minimum score = 0, maximum score = 10)
Itching | From baseline to visit 3 (40 days after the start of the treatment)
  Visual analogue scale (VAS) (minimum score = 0, maximum score = 10)
Epithelialization | From baseline to visit 3 (40 days after the start of the treatment)
  The degree of epithelialization of the fissure was determined at each visit and stratified using 3 levels (1 to 3) corresponding to <50%, >50% of healing or complete healing, respectively.
Physical and mental health | From baseline to visit 3 (40 days after the start of the treatment)
  Short-Form 12 (SF-12)
Physical and mental health | At visit 3 (40 days after the start of the treatment)
  SF-36 - Physical component score (PCS)
Physical and mental health | At visit 3 (40 days after the start of the treatment)
  SF-36 - Mental component score (MCS)
Patients' satisfaction | At visit 3 (40 days after the start of the treatment)
  VAS (1 = unsatisfied; 2 = neutral; 3 = quite satisfied; 4 = very satisfied; 5 = extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Hospital Treviso, Treviso, Italy

IPD SHARING:
Plan to Share IPD: No